CLINICAL TRIAL: NCT00810940
Title: Phase 1/2 Multicenter, Randomized, Controlled Trial of ABELADRUG200 in Closed, Severe Head Injury
Brief Title: Controlled Trial of ABELADRUG200 in Closed, Severe Head Injury
Acronym: ABELADRUG200
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abela Pharmaceuticals, Inc. (Industry)
Collaborators: Ohio State University (Other); University of California, Irvine (Other); Dr. Mahajan's Hospital & Industrial Trauma Centre (Other)
Responsible Party: Colette Cozean, Ph.D., CEO, Abela Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbelaTBI2
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Severe Head Trauma
Keywords: TBI; closed head injury; severe head trauma; traumatic brain injury
MeSH Terms: conditions — Craniocerebral Trauma; Head Injuries, Closed; Brain Injuries, Traumatic | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Control: Standard treatment for severe head trauma including mannitol
  Interventions: Drug: mannitol
- 2 (Experimental): Study drug plus standard treatment
  Interventions: Drug: AbelaDrug200

INTERVENTIONS:
Drug: AbelaDrug200 — IV 200 ml 28%drug in D5W every six hours, 10 min. duration, until ICP < 20 mmHg, then IV 100 ml same schedule for 24 hours
  Arms: 2
Drug: mannitol — mannitol plus standard treatment
  Arms: 1

SUMMARY:
This is a randomized, controlled clinical trial at three sites to determine the safety and preliminary efficacy of the study drug to treat severe head trauma (GCS 4-8). It is hypothesized that the drug may lower pressure in the brain, reduce mortality and the patient may have improved neurological function following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis TBI
* GCS 4-8
* Age 16-70

Exclusion Criteria:

* Multiple trauma resulting in shock
* Bilateral absent pupil response
* Time from injury > 6 hours
* Brain tumor or mass effect secondary to hemorrhage or brain surgery
* Pregnancy
* Confounding condition or injury
* Spinal cord injury
* Sustained high blood pressure or arterial oxygen saturation

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
reduction in intracranial pressure | 24 hours, 5 days

SECONDARY OUTCOMES:
mortality | 3 months
Glasgow Outcome Scale | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Boston University Medical Center, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio